CLINICAL TRIAL: NCT03362645
Title: Diagnostic Value of the Electrocardiogram in Fabry Disease
Acronym: DEFY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 16-005
Record Dates: First submitted 2016-08-29; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Fabry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fabry cardiomyopathy
- Hypertrophic cardiomyopathy

SUMMARY:
Cardiac complications occur in 78% of patients with Fabry disease and are mainly characterized by a high frequency of left ventricular hypertrophy resulting from an accumulation of GL3 in cardiomyocytes. Apart from family screening, left ventricular hypertrophy is an important factor in the diagnosis of Fabry disease. This left ventricular hypertrophy is more often concentric and homogeneous, but it can also be asymmetric and mimic the patterns seen in so-called familial hypertrophic cardiomyopathies caused by mutations in the sarcomere protein genes. Electrocardiogram has been suggested as a screening tool for Fabry disease. Analysis of the PQ interval would be of interest. An algorithm has even been proposed to differentiate Fabry disease from amyloidosis with excellent sensitivity and specificity. The only criterion of left ventricular hypertrophy used in all studies is the Sokolov-Lyon index, but this index has many limitations and does not appear to be discriminatory for Fabry disease. Other validated criteria for left ventricular hypertrophy, such as the Cornell, Lewis, Gubner index or the Romhilt-Estes point score, have never been tested in Fabry disease. The primary objective of our study is to evaluate the diagnostic value of different electrocardiographic scores of left ventricular hypertrophy in Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years, with genetically confirmed Fabry disease complicated by LVH.
* Patients aged > 18 years, with sarcomeric hypertrophic cardiomyopathy.

Exclusion Criteria:

* Patients aged < 18 years. Sarcomeric hypertrophic cardiomyopathy for which Fabry disease has not been excluded by alpha-galactosidase A assay (in men) and genetic analysis (GLA gene mutation) in women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 18 years, with genetically confirmed Fabry disease complicated by LVH.
  Patients aged > 18 years, with sarcomeric hypertrophic cardiomyopathy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Analysis of the PQ interval with a new algorithm | baseline
  Determine whether electrocardiographic criteria of left ventricular hypertrophy allow to distinguish between Fabry disease and sarcomeric hypertrophic cardiomyopathy